CLINICAL TRIAL: NCT00137800
Title: A Phase II Study of OSI-774 (Tarceva) in Elderly Subjects With Previously Untreated Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of OSI-774 (Tarceva) in Previously Untreated Elderly Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Pasi A. Janne, MD, PhD, Associate Professor, Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-308
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non-Small Cell Lung Cancer; Elderly Cancer Patients; Tarceva; Erlotinib; OSI-774; Stage IIIB or IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tarceva (Experimental): Chemotherapy Single Agent Systemic
  Interventions: Drug: OSI-774 (Tarceva)

INTERVENTIONS:
Drug: OSI-774 (Tarceva) — Once daily without interruption as long as there is no disease progression or serious side effects experienced.

SUMMARY:
The primary purpose of this study is to determine whether the drug OSI-774 is less toxic and potentially as good as or better than standard chemotherapy drugs, when given to subjects with non-small cell lung cancer, who are 70 years of age or older.

DETAILED DESCRIPTION:
Patients will receive OSI-774 once daily without interruption. There are no pre-determined number of cycles or planned dose interruptions. For the purposes of evaluation, toxicity and efficacy, a four week (28 day period) will be considered 1 cycle.

Patients will continue to receive OSI-774 until they develop progressive disease, unacceptable side-effects or wish to withdraw from the study.

Patients will have radiographic evaluations after every two cycles of therapy. After cycle 2, patients will also be evaluated by FDG-PET scanning.

Patients will also be asked to fill out a Lung Cancer Symptom Scale (LCSS) on the first day of each cycle.

Bloodwork will also be performed on day 1 of each cycle as well as at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 70 years of age or older
* Stage IV or IIIB non-small cell lung cancer (NSCLC)
* Measurable tumor(s)
* Three or more weeks since prior radiation therapy
* Three or more weeks since prior major surgery
* Must at least be able to walk and capable of taking care of oneself although unable to carry out work activities.
* Must be up and about more than 50% of waking hours.
* Life expectancy of 8 weeks or more
* Blood tests that show kidneys, liver and bone marrow to be working adequately
* Completely healed from previous oncologic or other major surgery

Exclusion Criteria:

* Prior chemotherapy regimen for non-small cell lung cancer
* Prior exposure to OSI-774 or similar treatments such as trastuzumab, ZD1839, C225, etc.
* Uncontrolled central nervous system metastases
* Concurrent active cancer
* Malignancies within the past 5 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Prior chemotherapy for any malignant disease
* Difficulty swallowing
* A disease or disorder that interferes with ability to digest and absorb food
* A medical condition that could make it unsafe for patient to participate in this study

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2005-05 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine how well non-small cell lung cancer cells in the body respond to OSI-774 | 2 years
To determine the survival rate of patients treated with OSI-774

SECONDARY OUTCOMES:
To determine the safety of OSI-774 in people 70 years of age or older | 2 years
To see how OSI-774 affects overall quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Janne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Perez-Soler R, Chachoua A, Hammond LA, Rowinsky EK, Huberman M, Karp D, Rigas J, Clark GM, Santabarbara P, Bonomi P. Determinants of tumor response and survival with erlotinib in patients with non--small-cell lung cancer. J Clin Oncol. 2004 Aug 15;22(16):3238-47. doi: 10.1200/JCO.2004.11.057. PMID 15310767
- See also: Dana-Farber Cancer Institute Lowe Thoracic Oncology Program — https://www.dana-farber.org/thoracic-lung-cancer-treatment-center/